CLINICAL TRIAL: NCT01145703
Title: Effects of Vitamin D Supplementation With and With Out Exercise on Metabolic and Physical Consequences of Vitamin D Deficiency in the Elderly
Brief Title: Vitamin D Supplementation and Metabolism in Vitamin D Deficient Elderly
Acronym: VitD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator terminated study due to low enrollment of eligible subjects
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute on Aging (NIA) (NIH); Nutrition Obesity Research Center (Other)
Responsible Party: Principal Investigator, Andrew P. Goldberg, GRECC Director, Professor of Medicine, Baltimore VA Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HP-00040570; P30AG028747 (NIH)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Vitamin D Deficiency; Metabolic Syndrome
Keywords: Body Composition; Cardiovascular Risk; Cognitive Function
MeSH Terms: conditions — Vitamin D Deficiency; Metabolic Syndrome | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RDA Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: RDA Vitamin D3 only
- Vit D repletion + 6M Supplementation (Experimental)
  Interventions: Dietary Supplement: Vitamin D2/3 Repletion only
- Vit D repletion + 6M Supplementation +AEX (Experimental)
  Interventions: Other: Vitamin D2/3 Repletion + AEX
- Vit D repletion + 6M Supplementation +RT (Experimental)
  Interventions: Other: Vitamin D2/3 Repletion + RT

INTERVENTIONS:
Dietary Supplement: RDA Vitamin D3 only — 800 IU of Vitamin D3 daily for 6 months
  Other Names: ergocalciferol
  Arms: RDA Vitamin D
Dietary Supplement: Vitamin D2/3 Repletion only — Vitamin D repletion with 50,000 IU of Vitamin D2/3 up to 3 x week(until levels are >75 nmol/l; 6-12wks) followed by 6 months maintenance supplementation with 2000 IU Vitamin D3 and up to 1000mg Calcium daily
  Other Names: cholecalciferol; ergocalciferol
  Arms: Vit D repletion + 6M Supplementation
Other: Vitamin D2/3 Repletion + AEX — Vitamin D repletion with 50,000 IU of Vitamin D2/3 up to 3 x week(until levels are >75 nmol/l; 6-12wks) followed by 6 months maintenance supplementation with 2000 IU Vitamin D3 and up to 1000mg Calcium daily plus aerobic exercise training
  Other Names: cholecalciferol; ergocalciferol
  Arms: Vit D repletion + 6M Supplementation +AEX
Other: Vitamin D2/3 Repletion + RT — Vitamin D repletion with 50,000 IU of Vitamin D2/3 up to 3 x week(until levels are >75 nmol/l; 6-12wks) followed by 6 months maintenance supplementation with 2000 IU Vitamin D3 and up to 1000mg Calcium daily plus resistance training
  Other Names: cholecalciferol; ergocalciferol
  Arms: Vit D repletion + 6M Supplementation +RT

SUMMARY:
The purpose of this study is to examine the effects of Vitamin D supplementation on the reasons (mechanisms) underlying the development of type 2 diabetes, metabolic syndrome (high blood pressure, cholesterol, diabetes, body weight/obesity), muscle weakness and wasting (sarcopenia), and impaired physical function (poor balance and walking) associated with vitamin D deficiency and osteopenia/osteoporosis (bone loss). The investigators obtain vitamin D through our diet and sunlight, and its conversion to active vitamins in the liver and kidneys promotes the intestinal absorption of calcium and regulation of bone growth. Therefore, vitamin D deficiency has been known for years to lead to weakened bones (osteopenia and osteoporosis). However, more recently, studies show vitamin D deficiency is associated with a number of other diseases, including type 2 diabetes, muscle weakness, frailty, and the metabolic syndrome. It has also been associated with cognitive impairment. Diabetes affects multiple organ systems including the heart, kidneys, musculoskeletal and nervous system. The possibility that vitamin D deficiency is linked to the development of type 2 diabetes, metabolic syndrome, muscle weakness and wasting (sarcopenia) and osteopenia/osteoporosis, and that vitamin D supplementation decreases the risk for these diseases, provides a relatively easy/accessible and inexpensive model of preventive therapy to decrease the incidence of these diseases. In addition, it is likely that genetic (inherited) factors play a role, but the relationship of these genes to these metabolic abnormalities have not been elucidated. Understanding the role of Vitamin D in health will allow us to translate these findings into therapy.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 years of age
* Women must be post menopausal (absence of menses for 12 months or greater)
* 25-hydroxyvitamin D level below 20 ng/ml (50 nmol/L)
* BMI 25-45 kg/m2
* Non smoker ( non smoking for at least 12 months:cigarettes, cigars, pipes)

Exclusion Criteria:

* Symptomatic heart disease, CAD, CHF, or uncontrolled hypertension (BP over 180 mm HG) unless medically stabilized
* Currently being treated for active cancer
* Type 1 diabetes; insulin treatment for diabetes, poorly controlled diabetes, HgA1c >10%
* Allergic to lidocaine
* History of seizures or taking anti-seizure or anti convulsion medications
* Untreated dyslipidemia with National Cholesterol ATPIII 10 year cardiac risk score greater than 10% (www.nhlbi.nih.gov/guidelines/cholesterol/atp3upd04.htm)
* Taking oral steroids, warfarin or other medications interfering with fat/muscle metabolism that may not be safely discontinued temporarily for specific procedures (ie for 72 hours prior)
* Taking medication that interfere with ability to replete Vitamin D
* Abnormal liver function 2 times normal levels
* Abnormal renal function (BUN above 40 mg/dl, Cr above 1.8 mg/dl, CrCl<60mg/dl)
* Hypercalcemia (Ca>10.2mg/dl)
* Anemia HCT below 30 mg/dl, platelets below 100,000/cm3
* Chronic pulmonary disease (on supplemental O2)
* Other systemic disorders that are not medically treated and stable or affect the ability to absorb Vitamin D.
* MMSE below 24, dementia or unstable clinical depression by exam
* Abnormal response to exercise test (ST segment depression greater than 2mm, chest pain, significant arrhythmias, extreme shortness of breath, cyanosis, exercising BP above 240/120 mm HG, or other contraindications to exercise) *requires follow up treatment w/ primary MD for continued participation in study
* Aerobically trained with VO2max greater than 2 SD above age-adjusted mean
* Participant is, in the opinion of the investigator, unable to adhere to the study protocol due to medical or orthopedic conditions that limit ability to exercise or travel to the Baltimore VA for protocol procedures.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
glucose tolerance and insulin sensitivity | Baseline, 3 months and 6 months

SECONDARY OUTCOMES:
muscle structure, inflammation and metabolic function to cause sarcopenia and frailty | Baseline, 3 months and 6 months
physical performance, balance and strength to increase strength and balance to reduce fall risk in older people | Baseline, 3 months and 6 months
cognitive function | Baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Goldberg, M.D., Principal Investigator — Baltimore VAMC/GRECC
Locations (1):
- Baltimore VAMC, Baltimore, Maryland, United States